CLINICAL TRIAL: NCT00779441
Title: An Open Label, Relative Bioavailability Study of 10 mg Zolpidem Tablet Under Non-Fasting Conditions
Brief Title: Bioequivalence Study of Zolpidem 10 mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif monif, Ranbaxy Research labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R05-275
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence zolpidem 10mg tablets
MeSH Terms: interventions — Zolpidem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Zolpidem 10mg tablets of ranbaxy
  Interventions: Drug: Zolpidem 10mg tablets
- 2 (Active Comparator): AmbienÂ® 10mg tablets
  Interventions: Drug: Zolpidem 10mg tablets

INTERVENTIONS:
Drug: Zolpidem 10mg tablets

SUMMARY:
The study compared the relative bioavailability (rate and extent of absorption) of 10 mg Zolpidem tablets by Ohm Laboratories Inc. with that of 10 mg AmbienÂ® tablets distributed by Sanofi-Synthelabo, Inc. following single oral dose (1x10 mg tablet) in healthy adult volunteers administered under non-fasting conditions

DETAILED DESCRIPTION:
This was a single-center, randomized, open label, two-way cross over study conducted under non-fasting conditions. Subjects checked into the clinical facility the day prior to dosing at least 10 hours prior to dose administration. On study day 1, subjects were dosed with single oral dose (1x10mg tablet) of the test and reference products thirty minutes after initiation of a standardized, high fat breakfast which was preceded by an overnight fast. Following a seven day wash out period, subjects returned and were dosed with an alternative treatment as per randomization Thirty-six (N=36) volunteers were enrolled in the study of which 17 were females and 19 were males. Subject 22 was dropped from further study participation prior to period II check in due to adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men or women 18 years of age or older at the time of dosing
2. Weights within Â±20% for height and body frame as per Desirable weight for adults(1983 Metropolitan Height and Weight table)
3. Volunteers judged by the investigator to be healthy based on their medical and medication history, physical examination, electrocardiogram, and clinical laboratory results
4. Volunteers willing to participate in the study and have signed a copy of written consent form
5. If female:

Of childbearing potential, was practicing an acceptable method of birth control for the duration of study as judged b y the investigator(s), such as condom with spermicide, intrauterine device (IUD), or abstinence; or Was menopausal for at least 1year; or Was surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

Subject candidates must not be enrolled in the study if they meet any of the following criteria:

1. Volunteers with a recent history of drug or alcohol addiction or abuse
2. Volunteers with the presence of clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators)
3. Volunteers with clinical laboratory test values outside the accepted reference range and, when confirmed on re-examination, were deemed to by clinically significant
4. Volunteers with a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody
5. Volunteers with positive drug abuse screen when screened for the study
6. Female volunteers demonstrating a positive pregnancy screen
7. Female volunteers who are currently breast feeding
8. Volunteers with a history of clinically significant allergies including the allergies
9. Volunteers with any clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigation)
10. Volunteers who currently use tobacco products
11. Volunteers who had taken any drug known to induce metabolism or inhibit hepatic metabolism in the 28 days prior to the period I dosing.
12. Volunteers who reported donating greater than 150 mL of blood within 28 days prior to period I dosing. All subjects were advised not to donate plasma for four weeks after completing the study
13. Volunteers who had donated plasma (e.g. plasmapheresis) within 14 days prior to period I dosing. All subjects were advised not to donate plasma for four weeks after completing o the study
14. Volunteers who reported receiving any investigational drug within 28 days prior to period I dosing
15. Volunteers who reported taking any systemic prescription 14 days prior to Period I dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-08; Primary Completion 2005-09 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html